CLINICAL TRIAL: NCT01500785
Title: Intracoronary Administration of Levosimendan in Cardiac Surgery Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Change of schedule
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCA-2011-1-3; 2011-002643-10 (EudraCT Number)
Record Dates: First submitted 2011-12-22; First posted 2011-12-28 (Estimated); Last update posted 2019-09-13 (Actual); Status verified 2019-09

CONDITIONS: Myocardial Stunning
MeSH Terms: conditions — Myocardial Stunning | interventions — Simendan; Vitamin B 12

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- levosimendan (Active Comparator)
  Interventions: Drug: levosimendan
- placebo (Placebo Comparator)
  Interventions: Drug: Vitamin B 12

INTERVENTIONS:
Drug: levosimendan — infusion; levosimendan (12 μg/kg) The study drug will be administered together with the induction of cardioplegia solution during five minutes (=once for each patient)
  Other Names: Simdax (manufacturer: Orion Corporation); CO1CX08
  Arms: levosimendan
Drug: Vitamin B 12 — Infusion made of Glucos B.Braun 50 mg/ml infusion together with vitamin B12 which is used to colour the glucose infusion to look identical to Simdax infusion The placebo will be administered together with the induction of cardioplegia solution during five minutes (=once for each patient).
  Other Names: Soluvit (B05XC)
  Arms: placebo

SUMMARY:
Incomplete recovery from ischemia causes stunned myocardium. Ischemia may be due to coronary artery disease or aortic cross-clamping during surgery. Stunning leads to myocardial dysfunction. It has been suggested that the mechanism responsible for the contractile depression in stunned myocardium is a decreased sensitivity of the myofibrils to calcium. Levosimendan is a calcium sensitizer, which has been shown to improve the function of stunned myocardium without obvious impairment of diastolic function. Systemic vasodilation and need of vasoconstrictive medication is usually apparent after administration of levosimendan. Colucci et al have demonstrated that with intracoronary administration of milrinone, another inodilator, systemic vasodilation could be excluded. If this is true with levosimendan, it may be possible to improve left ventricular hypo/dyskinesia without afterload reduction by adding levosimendan into cardioplegia solution.

The investigators hypotize that levosimendan, delivered together with cardioplegia, can improve LV dysfunction after opening of aortic cross-clamp in patients undergoing aortic valve and coronary artery bypass operation. Our primary endpoint is a change in cardiac output 15 min after separation from cardiopulmonary bypass compared to the baseline. Secondary endpoints are a change in LV ejection fraction from baseline to 5 min after sternal closure and cTnT/CK-MB on the first postoperative morning.

ELIGIBILITY:
Inclusion Criteria:

* preoperative LVEF 40% or less
* septal wall thickness more than 11mm
* less than moderate aortic insufficiency
* sinus rhythm before CPB

Exclusion Criteria:

* oesophageal disease
* known allergy to levosimendan or its metabolites or adjuvants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2019-09-11 (Actual)

PRIMARY OUTCOMES:
change in cardiac output | from baseline to 15min after weaning from CPB
  Our primary endpoint is a change in cardiac output 15 min after separation from cardiopulmonary bypass compared to the baseline (after induction of anesthesia).

SECONDARY OUTCOMES:
EF | from baseline to 5 min after sternal closure
  Secondary endpoint is a change in LV ejection fraction (EF) from baseline (after induction of anesthesia) to 5 min after sternal closure.
cTnT/CK-MB on the first postoperative morning. | from baseline to 1st post. op. morning
  Secondary endpoint is a change in cTnT/CK-MB on the first postoperative morning.

CONTACTS AND LOCATIONS:
Overall Officials: Panu Virkkala, MD, Principal Investigator — Heart Center Co. Tampere university hospital
Locations (1):
- Heart Center Co. Tampere university hospital, Tampere, Finland